CLINICAL TRIAL: NCT00117845
Title: Phase II Study of the Efficacy and Toxicity of Ontak (Denileukin Diftitox) in the Therapy of Adult T-Cell Leukemia
Brief Title: Phase II Study of the Efficacy and Toxicity of Ontak(Registered Trademark) (Denileukin Diftitox) in the Therapy of Adult T-Cell Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature closure as study drug is no longer available from the manufacturer.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Waldmann, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050185; 05-C-0185; NCT00138190 (obsolete NCT alias)
Record Dates: First submitted 2005-07-07; First posted 2005-07-08 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Leukemia, Adult T-Cell
Keywords: Denileukin Diftitox (Ontak); Recombinant Immunotoxin; Human T-Cell Lymphotropic Virus (HTLV1); CD25 Positive; IL-2R; ATL; Ontak; Adult T-Cell Leukemia; Lymphoproliferative Disorders
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Lymphoproliferative Disorders | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Denileukin Diftitox in ATL (Experimental): Denileukin Diftitox in adult T-cell leukemia (ATL) Patients will be treated with Denileukin Diftitox 9 mcg/kg/d intravenously for 5 days every 2 weeks.
  Interventions: Biological: Denileukin diftitox (Ontak)

INTERVENTIONS:
Biological: Denileukin diftitox (Ontak) — Patients will be treated with Denileukin Diftitox 9 mcg/kg/d intravenously for 5 days every 2 weeks.

SUMMARY:
Adult T-cell leukemia (ATL) is and aggressive characterized by the presence of cluster of differentiation 4 (CD4)/cluster of differentiation 25 (CD25)-expressing T cells (interleukin-2 [IL-2]R expressing) in the peripheral blood and in lymphoid and other tissues. Denileukin diftitox (Ontak(Registered Trademark)) is a genetically engineered fusion protein that targets IL-2-expressing malignancies. Denileukin diftitox interacts with the IL-2R on the cell surface, is internalized via endocytosis, and inhibits cellular protein synthesis, resulting in cell death within hours to days. The objectives of this study are to determine the clinical response to Denileukin diftitox of patients with adult T-cell leukemia (ATL) and the safety of Denileukin diftitox in those patients.

Eligible participants must be 18 years of age or older with chronic, lymphomatous and acute forms of ATL, and must be infected with human T-cell lymphotropic virus type I (HTLV1).

Patients will be treated with 9 mcg/kg/d of Denileukin diftitox intravenously for 5 days every 2 weeks. Tumor response will be evaluated after two cycles of treatment. Stable or responding patients will continue treatment for a total of 12 months, with evaluations every four cycles of treatment. Patients will be treated for two cycles beyond a complete remission. The trial uses an optimal two-stage design targeting for a true response proportion of more than 30 percent. Nine patients will be treated initially, with expansion to 29 patients if a response is seen in 1 of the initial 9 patients treated. Treatment will be discontinued if a patient experiences serious side effects.

A potential benefit is that a patient may undergo partial or complete remission. The research may not directly benefit participants, but the results may aid in the treatment of others.

DETAILED DESCRIPTION:
Background:

Adult T-Cell Leukemia is a lymphoproliferative disorder characterized by the presence of CD4/CD25 expressing T cells (IL-2R expressing) in the peripheral blood, in lymphoid and other tissues.

Denileukin diftitox is a genetically engineered fusion protein combining the enzymatically active domains of diphtheria toxin (DT) and the full length sequence of interleukin-2 (IL-2) that targets IL-2 expressing malignancies.

Denileukin diftitox interacts with the IL-2 R on the cell surface, is internalized via endocytosis, and inhibits cellular protein synthesis resulting in cell death within hours to days.

Objective:

Determine the clinical response to Denileukin diftitox (Ontak) of patients with adult T-cell leukemia (ATL).

Define the safety of Denileukin diftitox in patients who have ATL.

Eligibility:

Patients with chronic, lymphomatous and acute forms of ATL.

Patients must be human T-cell lymphotropic virus type I (HTLV1) positive.

Design:

Patients will be treated with 9mcg/kg/d of Denileukin diftitox for five days, on an every two week schedule.

Tumor response will be evaluated after two cycles of treatment. Stable or responding patients will continue treatment with evaluations every four cycles of treatment. Patients will be treated for two cycles beyond a complete remission.

The trial uses an optimal 2 stage design targeting for a true response proportion greater than 30%. Nine patients will be treated initially with expansion to 29 patients if a response is seen in one of the initial nine patients treated. If no response is seen at the 9 mcg/kg/d dose an additional 9 patients will be treated at a dose of 18 mcg/kg/d with expansion to 29 patients at this dose level if a response is seen. A stopping rule for excessive toxicity will be incorporated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have serum antibodies directed to human T-lymphotropic virus type 1 (HTLV-I).

All patients must have a histologically confirmed diagnosis of adult T-cell leukemia/lymphoma and more than 10% of the malignant cells must express cluster of differentiation 25 (CD25).

All stages of Tac-expressing adult T cell leukemia except smoldering are eligible: patients with chronic, lymphomatous or acute adult T-cell leukemia (ATL) are eligible. (See appendix 2 for characteristics of patients with the various stages of ATL)

Patients must have measurable disease. All patients with greater than 10% abnormal (i.e. TAC homogenous strongly expressing) peripheral blood mononuclear cells (PBMC) in the peripheral blood will be deemed to have measurable disease.

The patient must have a granulocyte count of at least 1000/mm^3 and a platelet count of greater than or equal to 50,000/mm^3.

Patients must have a creatinine of less than 2.0 mg/dl.

Omission of cytotoxic chemotherapy for ATL for 3 weeks prior to entry into the trial is required. However, patients receiving corticosteroids will be eligible.

Patients must have a life expectancy of greater than 2 months.

Eligible patients must be greater than or equal to 18 years old. There is no upper age limit.

Patients must have serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) value less than or equal to 2.5 times the upper limit of normal and bilirubin less than or equal to 3.0/dl. If a liver function test is judged to be elevated due to the underlying ATL, this parameter will be considered an unevaluable parameter for toxicity determinations.

Patients must have a serum albumin greater than or equal to 2.5 g/dl

Patients must be able to understand and sign an Informed Consent form.

All patients must use adequate contraception during participation in this trial and for three months after completing therapy.

EXCLUSION CRITERIA:

Patients with symptomatic leukemic meningitis will be excluded. However, patients that have both ATL and another HTLV-I-associated disease, tropical spastic paraparesis (TSP), will be included.

Pregnant and nursing patients are not eligible for the study.

Human immunodeficiency virus (HIV) positive patients are excluded from the study. Denileukin diftitox may produce a different pattern of toxicities in immunocompromised individuals.

Patients with Smoldering ATL are excluded.

Patients with serious intercurrent illnesses, past history of a myocardial infarction within 6 months or severe coronary artery disease

Patients who previously received Denileukin diftitox are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-07-11 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Waldmann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yates AD, Morgan WT, Watkins WM. Linkage-specific alpha-D-galactosidases from Trichomonas foetus: characterisation of the blood-group B-destroying enzyme as a 1, 3-alpha-galactosidase and the blood-group P1-destroying enzyme as a 1, 4-alpha-galactosidase. FEBS Lett. 1975 Dec 15;60(2):281-5. doi: 10.1016/0014-5793(75)80731-9. No abstract available. PMID 6322
- [Background] Uchiyama T, Yodoi J, Sagawa K, Takatsuki K, Uchino H. Adult T-cell leukemia: clinical and hematologic features of 16 cases. Blood. 1977 Sep;50(3):481-92. No abstract available. PMID 301762
- [Background] Poiesz BJ, Ruscetti FW, Gazdar AF, Bunn PA, Minna JD, Gallo RC. Detection and isolation of type C retrovirus particles from fresh and cultured lymphocytes of a patient with cutaneous T-cell lymphoma. Proc Natl Acad Sci U S A. 1980 Dec;77(12):7415-9. doi: 10.1073/pnas.77.12.7415. PMID 6261256
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0185.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denileukin Diftitox in ATL
Started | 17
Completed | 16
Not Completed | 1
Not completed — stopped treatment/drug supplyinterrupted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denileukin Diftitox in ATL
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.46 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate is based on the number of patients who achieve either a complete response (CR) or partial response (PR) to therapy. Complete response is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy and normalization of those biochemical abnormalities (for example LDH) definitely assignable to the lymphoma. Partial response is reduction by >=50% of leukemia cell count or >=50% reduction is the size of all measurable lesions, and no increase in size of any measurable or evaluable lesion or appearance of new lesion.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Denileukin Diftitox in ATL
Number analyzed (Participants) | 17
Participants
  Complete Response | 0
  Partial Response | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Denileukin Diftitox in ATL
Number analyzed (Participants) | 17
Participants | 17

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 72 months.
Arm/Group | Denileukin Diftitox in ATL
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denileukin Diftitox in ATL (N=17)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Obstruction/stenosis of airway::Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Perforation, GI::Duodenum (Gastrointestinal disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denileukin Diftitox in ATL (N=17)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 10 (39)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 12 (48)
Acute vascular leak syndrome (Vascular disorders) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12 (36)
Alkaline phosphatase (Metabolism and nutrition disorders) | 9 (20)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
Amylase (Metabolism and nutrition disorders) | 2 (6)
Anorexia (Gastrointestinal disorders) | 4 (4)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 (4)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (16)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 8 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (5)
Cardiac troponin I (cTnT) (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Creatinine (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 6 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (6)
Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 9 (27)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 5 (8)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 14 (44)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infection (Infections and infestations) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Colon
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Larynx
Infection (Infections and infestations) | 1 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Pharynx
Infection - Other (Specify, infection with neutropenia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 2 (3)
Insomnia (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (19)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 14 (56)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (5)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (10)
Metabolic/Laboratory - Other (Specify, hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 2 (2)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Neuropathy: cranial::CN I Smell (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (17)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 7 (9)
Pain - Other (Specify, Rt lumbar radiculopathy) (General disorders) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (3)
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 7 (9)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain::Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Tumor pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 (11)
Platelets (Blood and lymphatic system disorders) | 9 (13)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Proteinuria (Metabolism and nutrition disorders) | 4 (6)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other (Specify,) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — diminished SOB, fine crackles lower base, Pt states no SOB
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4)
Rigors/chills (General disorders) | 7 (10)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 (14)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 1 (2)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 7 (11)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (8)
Vomiting (Gastrointestinal disorders) | 7 (9)
Weight gain (General disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT00117845/Prot_SAP_000.pdf
  • Informed Consent Form (2011-06-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT00117845/ICF_001.pdf